CLINICAL TRIAL: NCT00753363
Title: Exercise, Inflammation and Pro-thrombotic Modulators in the Elderly
Brief Title: Exercise and Inflammation in the Elderly
Acronym: IRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Maryland (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AGCG-003-05F
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-03

CONDITIONS: Inflammation; Insulin Sensitivity
Keywords: Glucose Metabolism
MeSH Terms: conditions — Inflammation; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): 6 months of aerobic exercise training
  Interventions: Other: Aerobic Exercise Training
- Arm 2 (Experimental): 6 months of weight loss
  Interventions: Other: Weight Loss

INTERVENTIONS:
Other: Weight Loss — 6 months of weight loss
  Arms: Arm 2
Other: Aerobic Exercise Training — 6 months of aerobic exercise training
  Arms: Arm 1

SUMMARY:
Persistent low-grade inflammation and impaired fibrinolysis, are independent predictors of several chronic diseases highly prevalent in the older Veteran population including cardiovascular disease (CVD), stroke, and diabetes. Inflammation is likely to be a causative underlying mechanism of insulin resistance. Lifestyle changes such as weight loss and physical activity are advocated for the treatment of these chronic diseases and endpoints, and data are emerging which suggest that these treatments may be beneficial, in part, due to their anti-inflammatory effects. Identification of effective therapies that reduce chronic inflammation for Veterans is important given the widespread adverse health effects of a chronically elevated inflammatory state.

DETAILED DESCRIPTION:
This study will compare the effects of 6 month trial of aerobic exercise (AEX) vs. weight loss (WL) in older individuals on:

1. adipokine secretion and expression (tumor necrosis factor alpha, adiponectin);
2. adipose tissue and skeletal muscle inflammatory proximal receptor expression (adiponectin and tumor necrosis factor alpha expression) and signaling pathways; and
3. whether the changes in signal transduction are associated with changes in peripheral whole body insulin sensitivity by a hyperinsulinemic-euglycemic clamp.

The prevention and treatment of insulin resistance, the metabolic syndrome, and their CVD complications through exercise and weight loss could improve Veterans' health and reduce health care costs. Knowledge of their effectiveness has important implications for the cardiovascular health of Veterans given the widespread adverse health effects of chronic inflammation on vascular biology, skeletal muscle function and insulin action.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* 45-80 yrs of age
* Non-smoking for one year
* Body mass index greater than 20 kg/m2 and less than 50 kg/m2
* Menopause over 1 year

Exclusion Criteria:

* Symptomatic heart disease, coronary artery disease, congestive heart failure, or uncontrolled hypertension (blood pressure over 180/100 mm Hg) unless medically stabilized
* Currently being treated for active cancer
* Type 1 diabetes; Insulin or oral agent treatment for diabetes, poorly controlled diabetes fasting blood glucose over 160 mg/dl
* Allergic to lidocaine
* Untreated dyslipidemia with National Cholesterol Adult Treatment Panel III 10 year cardiac risk score greater than 10%, or receiving triglyceride lowering meds
* Other systemic disorders that are not medically treated and stable
* Taking beta-blockers, oral steroids, warfarin or any other medications interfering with fat/muscle metabolism that may not be safely discontinued temporarily for specific procedures (ie for 72 hours prior)
* Abnormal response to exercise test (ST segment depression greater than 2mm, chest pain, significant arrhythmias, extreme shortness of breath, cyanosis, exercising BP above 240/120mm Hg, or other contraindications to exercise) *requires follow up treatment w/ primary MD for continued participation in study
* Abnormal liver function
* Abnormal renal function
* Chronic pulmonary disease
* Anemia hematocrit below 35 mg/dl, platelets below 100,000/cm3
* Mini-mental state exam below 24, dementia or unstable clinical depression by exam
* Aerobically trained with maximal oxygen consumption greater than 2 standard deviations above age-adjusted mean
* Exercise group only: History of cerebrovascular disease (by medical history) with symptoms limiting the ability to exercise

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2012-11-29 (Actual); Study Completion 2012-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice S Ryan, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 59 | 60
Completed | 19 | 21
Not Completed | 40 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Customized [Mean (Full Range); unit: years]
  Age | 62 [45 to 81] | 61 [49 to 74] | 61 [45 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 19 | 20 | 39
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 32.4 (6.0) | 35.7 (4.4) | 34.1 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Insulin resistance is defined as a reduction in glucose utilization rate elicited by a given insulin concentration. Glucose utilization is measured during a three hour hyperinsulinemic-euglycemic clamp and is presented as a measure of insulin sensitivity. This is one of the most sophisticated methods to measure insulin sensitivity.
Time Frame: Baseline and 6 month
Measure: Mean (Standard Error); unit: μmol/kgFFM/min
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 19 | 21
μmol/kgFFM/min
  baseline | 50.2 (4.5) | 40.7 (6.2)
  6 month | 57.5 (4.9) | 42.3 (6.1)

2. Secondary Outcome: Body Weight
Time Frame: Baseline and 6 month
Measure: Mean (Standard Error); unit: kg
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 19 | 21
kg
  baseline | 93.3 (3.8) | 103.0 (3.9)
  6 month | 93.1 (4.2) | 93.7 (3.5)

3. Secondary Outcome: Fitness
Description: Maximal oxygen consumption (VO2max) on a treadmill
Time Frame: Baseline and 6 month
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 19 | 21
L/min
  Baseline | 2.38 (0.14) | 2.34 (0.12)
  6 month | 2.70 (0.15) | 2.29 (0.13)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between baseline and 6 months.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 0/59 | 1/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=59) | Arm 2 (N=60)
Dizzy and nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes